CLINICAL TRIAL: NCT02390856
Title: Randomized Controlled Trial: Volar Plate vs. Conventus DRS Intramedullary Fixation for Distal Radius Fractures
Brief Title: Volar Plate vs. Conventus DRS Fixation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Conventus Orthopaedics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-211
Record Dates: First submitted 2015-02-25; First posted 2015-03-18 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Fractures, Closed
MeSH Terms: conditions — Fractures, Closed

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Volar Plate (Active Comparator): Patients in this group will undergo distal radius fracture fixation with a traditional volar plate.
  Interventions: Device: Volar Plate
- Conventus DRS (Experimental): Patients in this group will undergo distal radius fracture fixation with the Conventus DRS intramedullary fixation device.
  Interventions: Device: Conventus DRS

INTERVENTIONS:
Device: Conventus DRS — The Conventus DRS (TM) is an intramedullary device intended to treat distal radius fractures. The device remains flexible during placement, but is made rigid at the completion of the surgical implant procedure. The implant is made from titanium alloy (Ti-6A1-4V) and Nitinol.
  Other Names: Conventus DRS Intramedullary Fixation Device
  Arms: Conventus DRS
Device: Volar Plate — A volar plate is a metallic plate fastened directly to the fractured bone with screws, to hold the fracture fragments in proper position. Volar plate fixation is the traditional surgical method for distal radius fractures.
  Arms: Volar Plate

SUMMARY:
Open reduction and internal fixation (ORIF) of unstable distal radius fractures is performed using a variety of fixation techniques. The most common method is fixed angle volar plate application. The investigators plan to compare the outcomes of fixed angle volar plating with a novel FDA approved intramedullary fixation device, Conventus DRS.

DETAILED DESCRIPTION:
Distal radius fractures are the most common fractures in the upper extremity. While a widely used method of fracture fixation, numerous studies have shown that locked volar plate fixation is associated with soft tissue irritation, flexor and extensor tendon rupture, and screw penetration of the radiocarpal or the distal radioulnar joint (DRUJ). Prominent hardware mandates hardware removal in 5-18% of cases.

Intramedullary fixation has recently received more attention in the literature because of the minimally invasive procedure required for device implantation. Additionally, because intramedullary fixation places the implant within the bone instead of onto it, the lack of implant exposure, as well as decreased soft tissue dissection, carries the potential for decreased inflammation at the surgical site. This prospective randomized case series will evaluate the clinical and functional outcomes of an expandable intramedullary fixation device and compare the complication profile with traditional fixed angle volar locked plating in a single-surgeon case series at a single hospital.

The wide variety of distal radius fractures demand customized treatment, and a number of different surgical treatments methods are available.(1) While percutaneous/external fixation, dorsal plating, fragment specific fixation, and intramedullary rod fixation have been studied, volar locked plate fixation has emerged over the past decade as the most common and versatile method of fracture fixation. Unfortunately, soft tissue and hardware complications continue to plague volar plate fixation, including digital stiffness, loss of forearm rotation, tendinopathy and tendon rupture, nerve injury and compression, hardware irritation, screw prominence, CRPS, and malunion.

Tarallo et al performed a retrospective review of 303 patients who had undergone volar plate fixation and found that implant-related complications had occurred in 5% of the patients (2). Of these, common complications seen were tendon rupture, screw loosening, and penetration into the articular space. While Tarallo et al studied only hardware related complications, other studies have reported complications associated of volar locking plate fixation as high as 22-27% (3,4). The flexor pollicis longus in particular is vulnerable to rupture, as hardware prominence at the watershed line of the distal radius exposes the FPL and other flexor tendons to frictional forces which result in fraying and rupture (5). Prominent pegs or screws dorsally threaten the extensor pollicis longus and neighboring extensor tendons.

Intramedullary fixation has limited data to date, and the current methods are applicable to a relatively narrow subset of radial fracture types. In a case series of three patients, Gunther and Lynch have shown that intramedullary fixation performed with a partially flexible rod that can be locked into rigid position once implanted in the bone resulted in good functional outcomes (6). Patients returned to their daily lives and at one-year post-operatively no adverse effects were reported. A prospective study analyzing the comparative functional outcomes between intramedullary nail versus volar plate fixation similarly found that functional recovery was comparative between the two groups, and that complication rates were slightly lower in the intramedullary fixation cohort (7). The authors of this study however noted the continued potential for screw penetration into the distal radioulnar joint (DRUJ).

The Conventus DRS expandable intramedullary fixation device used in this proposed study is FDA approved. A cadaveric study compared the fixation strength of the Conventus DRS with fixed angle volar plate fixation and demonstrated equivalency between the two for axial compression mean stiffness and dorsal bend mean stiffness (8). The Conventus DRS has been used in Europe where over 250 patients have been treated with the device. A safety and efficacy 'white paper' of the first 60 patients treated for a wide variety of fractures demonstrated excellent improvements in DASH scores with few hardware related events and an overall adverse event profile of 8.3%. (9) There was one re-operation for loss of fixation and four minor cases of neuritis that resolved. The device is FDA-approved in the US, and is being used across the country.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature patients (18-80)
* Unstable AO Type A and C1 fractures
* Closed injuries, acute (<14 days), displaced, and unstable

Exclusion Criteria:

* Patients under the age of 18 or over the age of 85 (if included in our analysis, these would likely be outliers in our patient population)
* Patients with documented complex regional pain syndrome (CRPS) or history of CRPS
* Patients with suspected or known allergies to titanium or nickel
* Patients who are non-English speakers
* Patients with open wound fractures
* Patients with inflammatory arthritis
* Patients with positive pregnancy test
* Additional musculo-skeletal injuries of the upper extremity would represent exclusion criteria (elbow fractures, scaphoid fractures, and contralateral wrist fracture).
* Previous major wrist injury or surgery (not including Carpal Tunnel, De Quervain's and trigger finger release)
* Patients with previously diagnosed metabolic bone disease, currently being treated.
* Non-English speaking patients (validated, translated questionnaires are not available)
* Patients needing ipsilateral concomitant operations that will have material impact on the study
* Patients with previous wrist fractures, prior wrist injury, stiffness, degenerative joint disease, or pain
* Previous minor surgery - for carpal tunnel, de Quervain's, ganglion, etc. - does not constitute exclusion criteria

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Complications at 2 weeks | 2 weeks
  Patients will be followed for up to one year after surgery to assess any complications which may develop. Complications will be defined as:
  * Stiffness (defined as inability to touch fingertips to distal palmar crease, OR 45 degrees or more loss of supination or pronation [compared to uninjured wrist], OR BOTH)
  * Loss of reduction
  * Hardware breakage
  * Hardware removal
  * Return to OR
  * Tendinopathy
  * Tendon rupture
  * Neuropathy
  * Superficial infection
  * Deep infection
  * Wound dehiscence
  * Incisional pain
  * Chronic Regional Pain Syndrome (CRPS)
  * None
Change from Baseline in Complications at 6 weeks | 6 weeks
  Patients will be followed for up to one year after surgery to assess any complications which may develop. Complications will be defined as:
  * Stiffness (defined as inability to touch fingertips to distal palmar crease, OR 45 degrees or more loss of supination or pronation [compared to uninjured wrist], OR BOTH)
  * Loss of reduction
  * Hardware breakage
  * Hardware removal
  * Return to OR
  * Tendinopathy
  * Tendon rupture
  * Neuropathy
  * Superficial infection
  * Deep infection
  * Wound dehiscence
  * Incisional pain
  * Chronic Regional Pain Syndrome (CRPS)
  * None
Change from Baseline in Complications at 3 months | 3 months
  Patients will be followed for up to one year after surgery to assess any complications which may develop. Complications will be defined as:
  * Stiffness (defined as inability to touch fingertips to distal palmar crease, OR 45 degrees or more loss of supination or pronation [compared to uninjured wrist], OR BOTH)
  * Loss of reduction
  * Hardware breakage
  * Hardware removal
  * Return to OR
  * Tendinopathy
  * Tendon rupture
  * Neuropathy
  * Superficial infection
  * Deep infection
  * Wound dehiscence
  * Incisional pain
  * Chronic Regional Pain Syndrome (CRPS)
  * None
Change from Baseline in Complications at 1 year | 1 year
  Patients will be followed for up to one year after surgery to assess any complications which may develop. Complications will be defined as:
  * Stiffness (defined as inability to touch fingertips to distal palmar crease, OR 45 degrees or more loss of supination or pronation [compared to uninjured wrist], OR BOTH)
  * Loss of reduction
  * Hardware breakage
  * Hardware removal
  * Return to OR
  * Tendinopathy
  * Tendon rupture
  * Neuropathy
  * Superficial infection
  * Deep infection
  * Wound dehiscence
  * Incisional pain
  * Chronic Regional Pain Syndrome (CRPS)
  * None

SECONDARY OUTCOMES:
Wrist Range of Motion | Up to 1 year
  Patients will be followed for up to one year after surgery to assess wrist motion (measurements of flexion, extension, radial deviation, ulnar deviation pronation, and supination)
Visual Analog Pain (VAS) Score | Up to 1 year
  VAS scores (0-10) will be obtained at standard clinical follow-up up to 1 year, after the scale of 0-10 (no pain - worst pain) has been explained
Patient-Rated Wrist Evaluation (PRWE) questionnaire | Up to 1 year
  The PRWE is a 15-item questionnaire designed to measure wrist pain and disability in activities of daily living. It will be administered at clinical follow-ups up to 1 year after surgery at 2 weeks, 6 weeks, 3 months, and 1 year postoperatively.
Tourniquet time | Time of Surgery
  On one occasion, on the day of surgery, tourniquet time will be recorded in minutes.
Operative time | Time of Surgery
  On one occasion, on the day of surgery, operative time will be recorded in minutes.
Articular Step off | Up to 1 year
  Articular step off will be assessed on x-rays at clinical follow-ups up to 1 year after surgery at 2 weeks, 6 weeks, 3 months, and 1 year postoperatively.
Articular Gap | Up to 1 year
  Articular gap will be assessed on x-rays at clinical follow-ups up to 1 year after surgery at 2 weeks, 6 weeks, 3 months, and 1 year postoperatively.
Volar tilt | Up to 1 year
  Volar tilt will be assessed on x-rays at clinical follow-ups up to 1 year after surgery at 2 weeks, 6 weeks, 3 months, and 1 year postoperatively.
Radial inclination | Up to 1 year
  Radial inclination will be assessed on x-rays at clinical follow-ups up to 1 year after surgery at 2 weeks, 6 weeks, 3 months, and 1 year postoperatively.
Ulnar variance | Up to 1 year
  Ulnar variance will be assessed on x-rays at clinical follow-ups up to 1 year after surgery at 2 weeks, 6 weeks, 3 months, and 1 year postoperatively.
Coronal Shift | Up to 1 year
  Coronal shift will be assessed on x-rays at clinical follow-ups up to 1 year after surgery at 2 weeks, 6 weeks, 3 months, and 1 year postoperatively.
Grip Strength | Up to 1 year
  Grip strength will be measured by the PI of the study with a Jamar grip dynamometer at clinical follow-ups up to 1 year after surgery at 2 weeks, 6 weeks, 3 months, and 1 year postoperatively.
Return to Work/Activities (quickDASH questionnaire) | Up to 1 year
  The QuickDASH is a shortened version of the DASH Outcome Measure. Instead of 30 items, the QuickDASH uses 11 items to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb. It will be administered at clinical follow-ups up to 1 year after surgery at 2 weeks, 6 weeks, 3 months, and 1 year postoperatively.
Pinch Strength | Up to 1 year
  Pinch strength will be measured by the PI with a Pinch Dynamometer at clinical follow-ups up to 1 year after surgery at 2 weeks, 6 weeks, 3 months, and 1 year postoperatively.
Intraoperative Complications | Time of Surgery
  Intraoperative complications will be assessed on 1 occasion, on the day of surgery. Intraoperative complications are defined as follows:
  * Loss of reduction
  * Conversion to alternate fixation
  * Hardware breakage
  * Fracture
  * Other
  * None

CONTACTS AND LOCATIONS:
Overall Officials: Scott W Wolfe, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Background] Tarallo L, Mugnai R, Zambianchi F, Adani R, Catani F. Volar plate fixation for the treatment of distal radius fractures: analysis of adverse events. J Orthop Trauma. 2013 Dec;27(12):740-5. doi: 10.1097/BOT.0b013e3182913fc5. PMID 23515129
- [Background] Rozental TD, Blazar PE. Functional outcome and complications after volar plating for dorsally displaced, unstable fractures of the distal radius. J Hand Surg Am. 2006 Mar;31(3):359-65. doi: 10.1016/j.jhsa.2005.10.010. PMID 16516728
- [Background] Arora R, Lutz M, Hennerbichler A, Krappinger D, Espen D, Gabl M. Complications following internal fixation of unstable distal radius fracture with a palmar locking-plate. J Orthop Trauma. 2007 May;21(5):316-22. doi: 10.1097/BOT.0b013e318059b993. PMID 17485996
- [Background] Limthongthang R, Bachoura A, Jacoby SM, Osterman AL. Distal radius volar locking plate design and associated vulnerability of the flexor pollicis longus. J Hand Surg Am. 2014 May;39(5):852-60. doi: 10.1016/j.jhsa.2014.01.038. Epub 2014 Mar 14. PMID 24630941
- [Background] Gunther SB, Lynch TL. Rigid internal fixation of displaced distal radius fractures. Orthopedics. 2014 Jan;37(1):e34-8. doi: 10.3928/01477447-20131219-14. PMID 24683654
- [Background] Gradl G, Mielsch N, Wendt M, Falk S, Mittlmeier T, Gierer P, Gradl G. Intramedullary nail versus volar plate fixation of extra-articular distal radius fractures. Two year results of a prospective randomized trial. Injury. 2014 Jan;45 Suppl 1:S3-8. doi: 10.1016/j.injury.2013.10.045. Epub 2013 Nov 4. PMID 24268189
- [Background] van Kampen RJ, Thoreson AR, Knutson NJ, Hale JE, Moran SL. Comparison of a new intramedullary scaffold to volar plating for treatment of distal radius fractures. J Orthop Trauma. 2013 Sep;27(9):535-41. doi: 10.1097/BOT.0b013e3182793df7. PMID 23187156
- [Background] Palmer AK, Hale JE. Conventus DRS Plating System: A Preliminary Report [White paper]. Conventus Orthopedics 2013. Retrieved from <http://www.conventusortho.com/wp-content/uploads/2015/03/4473-1-Rev-2-White-Paper-Conventus-Distal-Radius-System-A-Preliminary-Report.pdf>.